CLINICAL TRIAL: NCT02429986
Title: Observational and Transversal Study of Patients Treated in "Real Life"Conditions With Adaptive Servo-Ventilation
Brief Title: Adaptive Servo-Ventilation in "Real Life" Conditions : the OTRLASV Study
Acronym: OTRLASV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9498; 2014-A01565-42 (Other: RCB number)
Record Dates: First submitted 2015-04-01; First posted 2015-04-29 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Chronic Heart Failure and; Complex Sleep Apnea Syndrome; Obstructive Sleep Apnea Syndrome and; Idiopathic Central Sleep Apnea Syndrome; Idiopathic Induced Periodic Breathing; Central Sleep Apnea Syndrome
Keywords: Adaptive Servo-Ventilation; Chronic Heart Failure; Central Sleep Apnea Syndrome; Central and Obstructive Sleep Apnea Syndrome; Complex Sleep Apnea Syndrome; Hunter-Cheyne-Stokes Breathing; Periodic Breathing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASV Arm (Other): The measures are performed during the annual consultation required by the French Social Security for the renewal of the reimbursement of the ASV care.
  Interventions: Device: Adaptive Servo-Ventilation

INTERVENTIONS:
Device: Adaptive Servo-Ventilation — Adaptive Servo-Ventilation proceeds by continually measuring either minute ventilation or airflow and calculates a target ventilation to be applied as needed.

SUMMARY:
Adaptive Servo-Ventilation (ASV) treatment is routinely prescribed in France. In order to be reimbursed according to the French Social Security rules, the patient treated with an ASV needs to be examined each year. In this observational transversal single-visit study, the investigators aim to describe the clinical characteristics of patients treated with ASV and the associated device settings.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate in "real life conditions" the use of Adaptative Servo-Ventilation (ASV) treatment. ASV treatment is routinely prescribed in France in patients with various sleep disorders breathing (Chronic Heart Failure (CHF) and Central Sleep Apnea Syndrome (CSAS), CHF and central and obstructive sleep apnea (COSA), Obstructive Sleep Apnea Syndrome (OSAS) and complex sleep apnea syndrome (compSAS), idiopathic or drug induced periodic breathing.

In order to be reimbursed according to the French Social Security rules, the patient treated with an ASV needs to be examined each year. In this observational transversal single-visit study, the aim is to describe the clinical characteristics of patients treated with ASV and the associated device settings. The aim is to evaluate the safety and efficacy issues in real life conditions of the ASV prescription.Depending of the data, data are obtained after analysis of the six latest months data of the ASV device, after questioning the patient, after analysis of the polygraphy/oximetry (if prescribed by the doctor for the renewal consultation of the ASV care and reimbursement by the French Social Security). All the data are obtained during the annual consultation required by the French Social Security.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age more than 18 years (inclusive)
* Patient treated with ASV for at least one year,and eligible for care and for the reimbursement by the French Social Security rules.
* Patient presenting at the annual control consultation for the continuation of the ASV treatment according to the French Social Security rules.

Exclusion Criteria:

* Pregnancy, intention of being pregnant, breastfeeding.
* Inability to understand the nature and aims of the study or to communicate with the investigator
* Simultaneous participation in another trial with an exclusion clause to participate to an other trial.
* No affiliation to the French social security
* Loss of personal capacity resulting in state protection
* Deprivation of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Residual Apnea Hypopnea Index (AHI) evaluated by the ASV device and associated pressure settings | The measures are performed during the annual consultation required by the French Social Security for the renewal of the reimbursement of the ASV care. The measures are obtained after analysis of the six latest months data of the device.
  Relationship between the residual AHI and the associated pressure settings, in function of the phenotype of the patients (presence or absence of cardiopathy, presence or absence of altered left ventricular ejection fraction (≤45% or > 45%)

SECONDARY OUTCOMES:
Sleep Disorder Breathing involved in the initial prescription of ASV | The day of inclusion
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
ASV compliance (number of hour per day, number of day with ≥3 hours in the past 6 months) | The day of inclusion during the consultation or in a maximum delay of 15 days after (if the patient forgot to bring his device)
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Type of device used nad history of device used (CPAP used before ASV ?) | The day of inclusion during the consultation or in a maximum delay of 15 days after (if the patient forgot to bring his device)
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security)
Used or not of an auto-EPAP | The day of inclusion during the consultation or in a maximum delay of 15 days after (if the patient forgot to bring his device)
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Settings of the device (Inspiratory and Expiratory pressures, duration of pressurization, backup frequency) | The day of inclusion during the consultation or in a maximum delay of 15 days after (if the patient forgot to bring his device)
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Type of mask used and historical use of mask | The day of inclusion during the consultation or in a maximum delay of 15 days after (if the patient forgot to bring his device)
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Changes in AHI as compared to baseline | The day of inclusion during the consultation or in a maximum delay of 15 days after (if the patient forgot to bring his device)
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Changes in Daytime Sleepiness by measuring Epworth scale as compared to baseline if available | The day of inclusion
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Changes in Asthenia by measuring Pichot scale as compared to baseline if available | The day of inclusion
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Number of hospitalization during the last year and etiology of the hospitalization | The day of inclusion
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Presence of a cardiomyopathy | The day of inclusion
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Treatment of the cardiomyopathy (medication consumption and use of cardiac implant will be reported) | The day of inclusion
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).
Number of patients not showing up for the annual consultation | One year after the start of the study
  The data are obtained after questioning the patient (Epworth, Pichot and satisfaction scales) or after analysis of the six latest months data of the device or after analysis of the polygraphy/oximetry (if necessary and prescribed by the doctor in order to monitoring the patient for the renewal consultation of the ASV care and reimbursement by the French Social Security).

CONTACTS AND LOCATIONS:
Overall Officials: Dany JAFFUEL, MD, PhD, Principal Investigator — Polyclinic Saint-Privat
Locations (5):
- France (5):
  - Polyclinic Saint-Privat, Boujan-sur-Libron
  - CHU Dijon, Dijon
  - Hôpital Nord, Marseille
  - Arnaud de Villeneuve University Hospital, Montpellier
  - Hôpital Pitié Salpetrière, Paris

REFERENCES:
- [Result] Jaffuel D, Philippe C, Rabec C, Mallet JP, Georges M, Redolfi S, Palot A, Suehs CM, Nogue E, Molinari N, Bourdin A. What is the remaining status of adaptive servo-ventilation? The results of a real-life multicenter study (OTRLASV-study) : Adaptive servo-ventilation in real-life conditions. Respir Res. 2019 Oct 29;20(1):235. doi: 10.1186/s12931-019-1221-9. PMID 31665026
- [Result] Jaffuel D, Rabec C, Philippe C, Mallet JP, Georges M, Redolfi S, Palot A, Suehs CM, Nogue E, Molinari N, Bourdin A. Patterns of adaptive servo-ventilation settings in a real-life multicenter study: pay attention to volume! : Adaptive servo-ventilation settings in real-life conditions. Respir Res. 2020 Sep 21;21(1):243. doi: 10.1186/s12931-020-01509-7. PMID 32957983
- [Result] Jaffuel D, Mallet JP, Combes N, Palot A, Rabec C, Molinari N, Jaber S, Bourdin A. [Adaptive servo-ventilation after the SERVE-HF study: The swan song?]. Rev Mal Respir. 2016 Sep;33(7):641-4. doi: 10.1016/j.rmr.2016.04.001. Epub 2016 May 5. No abstract available. French. PMID 27155898